CLINICAL TRIAL: NCT05473026
Title: A Pilot Feasibility Study of a Gratitude Journaling Intervention to Enhance Well-being and Exercise Readiness in Older African American Female Breast Cancer Survivors
Brief Title: Grateful Strides Toward Physical Activity and Well-Being for Black Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB202201483; P30AG028740 (NIH)
Record Dates: First submitted 2022-07-13; First posted 2022-07-25 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cancer Survivors; African Americans; Women; Psychology, Positive; Cardiometabolic Syndrome; Exercise; Feasibility Studies; Breast Neoplasm Female
Keywords: African American Women; Breast Cancer Survivorship; Gratitude; Cardiometabolic Syndrome; Geriatrics; Physical Activity
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: Two-group parallel random-assignment experimental design.
Who Masked: Outcomes Assessor
Masking Description: The principal investigator will inform participants of their group assignment and provide intervention details. The research assistant and biostatistician will be blind to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gratitude Intervention (Experimental): Each participant will receive a gratitude journal (paperback or electronic journal based on preference) for eight weeks and will have the following journaling prompt to complete at least twice a week: "There are many things in our lives, both large and small, that we might be grateful about. Think back over the day and write down on the line below all that you are grateful for today" (maximum six reasons). The educational goal-setting component will be drawn from the American Cancer Society's Nutrition, Physical Activity, and Cancer toolkit. Participants will be able to choose the order in which they complete the goal-setting modules. Both exercises will be administered daily over eight weeks.
  Interventions: Behavioral: Gratitude Intervention
- Attention Control (No Intervention): Each participant will receive a journal (paperback or electronic journal based on preference) Participants will receive the following general journaling prompt to complete at least twice a week: "What are some memorable events that happened to you today, big, or small (maximum six memories). Write a brief statement about it.

INTERVENTIONS:
Behavioral: Gratitude Intervention — Gratitude journaling and goal setting for exercise readiness over eight weeks.
  Arms: Gratitude Intervention

SUMMARY:
This pilot study will assess the feasibility of a gratitude intervention to promote physical activity, and well-being and positively impact biomarkers of health among older African American breast cancer survivors. The intervention will also include a goal-setting component to promote exercise readiness and examine the cultural phenomena of the Superwoman schema among Black women.

DETAILED DESCRIPTION:
In this pilot feasibility study, the overall aims are:

Aim 1. Assess the feasibility and acceptability of a gratitude journaling intervention using a pilot randomized controlled trial (RCT) design over eight weeks. We hypothesize that among the 28 participants 1) at least 80% of the participants will report the intervention to be acceptable, 2) biomarker collection will be completed in at least 80% of the surveys and the retention rate will be 80% in each group, and 3) physical activity, health markers, gratitude, well-being, and distress will improve over time.

Aim 2. Describe distributions of outcome variables and effect size for the gratitude journaling intervention on dispositional gratitude, spiritual well-being, psychological distress, exercise readiness, mental and health behaviors in African American/Black women (Superwoman Schema), and inflammatory biomarkers from baseline to post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Self-report as AA or Black
* English speaking
* History of BC (Stage I-IV); 3 months to 6 years post-adjuvant chemotherapy
* Participants on hormonal therapies or HER-2 therapy are acceptable

Exclusion Criteria:

* Self-reported regular meditation or gratitude practices (more than once a week for at least a month)
* Meeting the CDC's physical activity guidelines (at least 150 min of moderate-intensity aerobic physical activity or 75 min of vigorous-intensity physical activity, or an equivalent combination each week)

Ages: 50 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakeshia Cousin, PhD, APRN, Principal Investigator — University of Florida
Locations (1):
- University of Florida CTSI Clinical Research Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cousin L, Braithwaite D, Anton S, Zhang Z, Lee JH, Leewenburgh C, Lyon D. A pilot study of a gratitude journaling intervention to enhance spiritual well-being and exercise self-efficacy in Black breast cancer survivors. BMC Psychiatry. 2024 Dec 18;24(1):931. doi: 10.1186/s12888-024-06362-2. PMID 39696111
- [Derived] Cousin L. Cardio-oncology disparities: Interplay of psychosocial stress, inflammation, and cardiometabolic health among Black breast cancer survivors. Am Heart J Plus. 2024 Jan 30;38:100366. doi: 10.1016/j.ahjo.2024.100366. eCollection 2024 Feb. PMID 38510748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited using organic social media recruitment, flyers, and multiple specialized strategies, including the OAIC Pepper Center Clinical Research Core - Participant Registry (IRB201601352), UF Health Cancer Center Community-Partnered Cancer Disparities Research Collaborative, UF Health Cancer Center Community Outreach and Engagement, UF Healthstreet, Integrated Data Repository, and UF Consent2Share Registries. Potential participants were screened for eligibility via telephone.
Period: Overall Study
Arm/Group | Gratitude Intervention | Attention Control
Started | 13 | 13
Completed | 8 | 11
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gratitude Intervention | Attention Control | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Demographics survey.
  years | 63.4 (6.5) | 66.7 (9.1) | 65.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Demographics survey.
  Participants
    Female | 13 | 13 | 26
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Demographics survey.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 13 | 13 | 26
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Demographics survey.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 13 | 13 | 26
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Demographics survey.
  kg/m2 | 36.1 (10.7) | 31.7 (5.7) | 33.9 (8.7)
Weight [Mean (Standard Deviation); unit: pounds] | 222.5 (69.3) | 181.1 (39.8) | 201.8 (59.3)
Height [Mean (Standard Deviation); unit: inches] — Demographics survey.
  inches | 65.5 (3.2) | 63.5 (2.8) | 64.5 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Met Inclusion Criteria Compared to Participants Approached
Description: Percentage of women who meet the inclusion criteria relative to the number of women approached.
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Gratitude Intervention | Attention Control
Number analyzed (Participants) | 13 | 13
Participants | 13 | 13

2. Primary Outcome: Participant Completion of Baseline Assessment Measures
Description: Percentage of participants completing baseline assessment measures.
Time Frame: Week 0
Measure: Count of Participants; unit: Participants
Arm/Group | Gratitude Intervention | Attention Control
Number analyzed (Participants) | 13 | 13
Participants | 13 | 13

3. Primary Outcome: Participant Completion of Both Baseline Assessments and Post-intervention Assessments
Description: Percentage of participants who completed baseline assessments and completed the post-intervention assessments.
Time Frame: Week 0, Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Gratitude Intervention | Attention Control
Number analyzed (Participants) | 13 | 13
Participants | 8 | 11

4. Primary Outcome: Treatment Satisfaction Using Client Satisfaction Questionnaire (CSQ-8)
Description: We assessed treatment satisfaction using the mean Client Satisfaction Questionnaire(CSQ-8) scores. An overall score is calculated by summing the respondent's rating score for each scale item. Scores range from 8 to 32, with higher values indicating higher satisfaction.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude Intervention | Attention Control
Number analyzed (Participants) | 13 | 13
score on a scale | 29.8 (3.7) | 29.2 (3.0)

5. Secondary Outcome: Change in Dispositional Gratitude From Baseline to Post-intervention
Description: The mean change of dispositional gratitude measured at week 0/baseline and post-intervention/week 8 was measured using the Gratitude Questionnaire-6 designed to measure four facets of dispositional gratitude: (a) intensity, (b) frequency, (c) span, and (d) density. The scale consists of six items, each rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). To calculate the GQ-6 score, each item's score is summed to yield a total score. The minimum possible score is 6, indicating the lowest level of gratitude, and the maximum possible score is 42, indicating the highest level of gratitude. For example, if a participant's responses to the six items are 5 (slightly agree), 6 (agree), 4 (neutral), 7 (strongly agree), 3 (slightly disagree), and 5 (slightly agree), the total score would be 30. This total score is then used to gauge the participant's level of gratitude, with higher scores reflecting greater gratitude.
Time Frame: Week 0, Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude Intervention | Attention Control
Number analyzed (Participants) | 13 | 13
score on a scale | 0.5 (1.3) | -0.3 (1.0)

6. Secondary Outcome: Change in Spiritual Well-being From Baseline to Post-intervention
Description: The Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being is a self-report measure designed to assess spiritual well-being in individuals with chronic illness. It was used to report mean change from week 0/baseline and post-intervention/week 8. The scale comprises 12 items divided into two subscales: Meaning/Peace and Faith. Each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). To calculate the FACIT-Sp-12 score, each item's score is summed. The Meaning/Peace subscale score is obtained by summing the scores of items 1 to 8, with a range of 0 to 32. The Faith subscale score is derived from items 9 to 12, with a range of 0 to 16. The total spiritual well-being score, which combines both subscales, ranges from 0 to 48. Higher scores on the FACIT-Sp-12 indicate greater spiritual well-being.
Time Frame: Week 0, Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude Intervention | Attention Control
Number analyzed (Participants) | 13 | 13
score on a scale | 3.6 (8.0) | -1.8 (3.1)

7. Secondary Outcome: Change in Distress From Baseline to Post-intervention
Description: The mean change of distress baseline/week 0 and post-intervention/week 8 was measured using the Perceived Stress Scale designed to measure stress during the last month. The scale consists of 10 items, each rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). To calculate the PSS score, each item's score is summed, with items 4, 5, 7, and 8 being reverse-scored to account for their positive phrasing. The reversed scoring for these items means that a response of 0 becomes 4, 1 becomes 3, 2 remains 2, 3 becomes 1, and 4 becomes 0. The total score, ranging from 0 to 40, reflects the individual's perceived stress level, with higher scores indicating greater stress.
Time Frame: Week 0, Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude Intervention | Attention Control
Number analyzed (Participants) | 13 | 13
score on a scale | -2.1 (4.9) | -1.3 (4.5)

8. Secondary Outcome: Change in Superwoman Schema (Racial and Gender Identity) From Baseline to Post-intervention
Description: The Giscombe Superwoman Schema Questionnaire (GSSQ) measured the mean change in Superwoman Schema between baseline and post-intervention at weeks 0 and 8. The GSSQ consists of 35 items across five dimensions: obligation to manifest strength (6 items), obligation to suppress emotions (7 items), resistance to being vulnerable (7 items), intense motivation to succeed (6 items), and obligation to help others (9 items). Items are rated on a Likert scale from 0 (not true) to 3 (true all the time). The total score ranges from 0 to 105, with subscale ranges as follows: Strength (0-18), Suppress (0-21), Resistance (0-21), Motivation (0-18), and Help (0-27). Higher scores indicate stronger endorsement of the Superwoman Schema. Total and subscale scores are summed, with higher scores representing stronger schema identification.
Time Frame: Week 0, Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude Intervention | Attention Control
Number analyzed (Participants) | 13 | 13
score on a scale
  Strength subscale | -0.4 (1.9) | -0.9 (3.9)
  Suppress emotions subscale | -0.8 (4.2) | 0.5 (5.2)
  Resistance to vulnerability subscale | -2.1 (4.2) | -0.3 (7.6)
  Motivation to succeed subscale | -1.3 (3.2) | -1.0 (4.4)
  Care for others subscale | 0.1 (5.5) | 1.3 (6.8)
  Total score | -4.4 (11.4) | 1.1 (23.9)

9. Secondary Outcome: Change in Exercise Readiness From Baseline to Post-intervention
Description: The Exercise Readiness Scale measured the stages of exercise behavior change at baseline and post-intervention. The scale consists of five items assessing exercise behavior and intentions. Participants choose one statement that best describes their current level of physical activity, with options ranging from 1 (no participation in physical activity and no intention to start) to 5 (exercising regularly for more than 6 months). Scores range from 1 to 5, with higher scores indicating greater readiness for regular physical activity and higher stages of exercise behavior change.
Time Frame: Week 0, Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude Intervention | Attention Control
Number analyzed (Participants) | 13 | 13
score on a scale | 0.8 (1.5) | -0.2 (0.6)

10. Secondary Outcome: Change in Tumor Necrosis Factor Alpha (TNF-α), Interleukin 6 (IL-6), Growth/Differentiation Factor-15 (GDF15) From Baseline to Post-intervention
Description: The mean change of inflammatory biomarkers baseline/week 0 and post-intervention/week 8 was measured using a Luminex panel containing Tumor Necrosis Factor Alpha (TNF-α), Interleukin 6 (IL-6), Growth/Differentiation Factor-15 (GDF15).
Time Frame: Week 0, Week 8
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Gratitude Intervention | Attention Control
Number analyzed (Participants) | 13 | 13
pg/mL
  TNF-a (pg/mL) | -2.4 (5.1) | -0.2 (1.1)
  IL-6 (pg/mL) | 3.0 (4.1) | 0.0 (15.3)
  GDF-15 (pg/mL) | 17.4 (89.4) | 15.2 (696.4)

11. Secondary Outcome: Change in C-Reactive Protein From Baseline to Post-intervention
Description: The mean change of inflammatory biomarkers baseline/week 0 and post-intervention/week 8 was measured using a Enzyme-linked immunosorbent assay (ELISA) kit containing C-Reactive Protein.
Time Frame: Week 0, Week 8
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Gratitude Intervention | Attention Control
Number analyzed (Participants) | 13 | 13
mg/L | 3.1 (6.0) | 0.6 (2.6)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Adverse events to subjects, if any, would have been recorded online in the form of the "Serious and Unexpected Adverse Event and Safety Report" developed by the University of Florida's IRB. This form collects a description of the event, the course of action taken, and specification regarding whether the event was: 1) serious (e.g., requiring hospitalization, resulting in significant disability/incapacity or death); 2) unexpected, and 3) more than likely related to the study procedures.
Arm/Group | Gratitude Intervention | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT05473026/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT05473026/ICF_000.pdf